CLINICAL TRIAL: NCT00037440
Title: Genetic Epidemiology of Change in CVD Risk Factors (HL70568-1)
Brief Title: Genetic Epidemiology of Change in CVD Risk Factors
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael Hallman, Assistant Professor, Epidemiology and Disease Control, The University of Texas Health Science Center, Houston
Other Study IDs: 1171; R01HL070568 (NIH)
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BHS Whites: Whites from Bogalusa, Louisiana; initially recruited as schoolchildren and followed at irregular intervals (about 3 years apart on average) into adolescence and early adulthood. There were no interventions of any kind-- this was an observational study only.
  Interventions: Genetic: Polymorphisms measured
- BHS African Americans: African Americans from Bogalusa, Louisiana, initially recruited as schoolchildren and followed at irregular intervals (about 3 years apart on average) into adolescence and early adulthood. There were no interventions of any kind-- this was an observational study only.
  Interventions: Genetic: Polymorphisms measured

INTERVENTIONS:
Genetic: Polymorphisms measured

SUMMARY:
To extend knowledge of the genetic factors affecting the course of cardiovascular disease risk factor development over a substantial portion of an individual's lifetime.

DETAILED DESCRIPTION:
BACKGROUND:

While the onset of symptomatic cardiovascular disease (CVD) typically occurs in middle age or later, the development of the underlying pathology is clearly a long-term process, and early-state lesions having been identified at autopsy even in children. Understanding the course of CVD risk development from childhood into middle age will clearly be valuable both in understanding the pathology of CVD and in targeting preventive measures most effectively. Furthermore, while genetic factors are agreed to play a significant role in the development of CVD, most genes contributing to interindividual variation in CVD risk will have relatively small effects on risk for any given individual, even though their aggregate effects contribute significantly to CVD risk in the overall population. Relatively little is known about the effects of genetic variants on the course of CVD risk factor development in individuals over time. The Bogalusa Heart Study (BHS), which began in 1973 as a study of CVD risk factors in children but evolved to cover the development of CVD risk factors from childhood into early middle age, offers an unparalleled resource for investigating the genetic factors influencing within-individual changes over time in quantitative factors, such as serum lipids and blood pressure, related to CVD risk.

DESIGN NARRATIVE:

Approximately 1500 individuals who were examined in the BHS on at least three separate occasions over a period of up to 20 years, and who consented to participate in studies of genetic factors influencing CVD risk, will have genotypes measured at selected loci either known or strongly suspected to affect interindividual variation in CVD risk. Longitudinal multilevel regression will be used to measure the effects of variation at these loci on quantitative CVD risk factor profiles within individuals and to determine whether some gene effects on CVD risk variation are age-dependent.

ELIGIBILITY:
Schoolchildren from Bogalusa, Louisiana. All children in Bogalusa public schools were eligible.

Ages: 8 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Community study of schoolchildren in Bogalusa, Louisiana, with follow-up into young adulthood. Both whites and African Americans recruited.
Sampling Method: Non-Probability Sample
Enrollment: 1735 (Actual)
Dates: Start 2001-09; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Plasma lipid levels | Change from 8 - 18 years of age

CONTACTS AND LOCATIONS:
Overall Officials: David Hallman, Principal Investigator — The University of Texas Health Science Center, Houston

REFERENCES:
- [Background] Hallman DM, Srinivasan SR, Chen W, Boerwinkle E, Berenson GS. The beta(2)-adrenergic receptor Arg16-gly polymorphism and interactions involving beta(2)- and beta(3)-adrenergic receptor polymorphisms are associated with variations in longitudinal serum lipid profiles: the Bogalusa Heart Study. Metabolism. 2004 Sep;53(9):1184-91. doi: 10.1016/j.metabol.2004.03.019. PMID 15334382